CLINICAL TRIAL: NCT07310433
Title: Dapagliflozin Combined With Next-generation Hormonal Agent (NHA) Versus Single NHA in Participants With Metastatic Castrate-resistant Prostate Cancer: a Phase 2, Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Dapagliflozin Combined With Next-generation Hormonal Agent (NHA) Versus Single NHA in Participants With Metastatic Castrate-resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yung NA (Other)
Collaborators: Ruijin Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Yung NA, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKURO202502
Record Dates: First submitted 2025-11-24; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer
Keywords: prostate cancer; sglt2
MeSH Terms: conditions — Prostatic Neoplasms | interventions — dapagliflozin; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): dapagliflozin 10 mg daily along with standard medical care (NHA + ADT)
  Interventions: Drug: Dapagliflozin (10mg Tab); Drug: standard medical care (ADT + NHA)
- Control (Active Comparator): Standard of Care (ADT + NHA)
  Interventions: Drug: standard medical care (ADT + NHA)

INTERVENTIONS:
Drug: Dapagliflozin (10mg Tab) — Dapagliflozin (10mg Tab)
  Arms: Intervention
Drug: standard medical care (ADT + NHA) — standard medical care for metastatic prostate cancer (ADT + NHA), the choice of NHA and ADT to be agreed among participant and treating physician with dosage and frequency according to local guideline. Surgical castration is also acceptable as ADT.

SUMMARY:
Dapagliflozin is a well-established medication being marketed and used for treatment Type 2 diabetes mellitus (T2DM). In retrospective cohort studies done by our team, we found that metastatic prostate cancer patients who received Dapagliflozin together with standard anti-cancer treatment, androgen deprivation therapy (ADT) combined with novel hormonal agent (NHA), had better tumor control than those having ADT and NHA.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) combined with novel hormonal agent (NHA) is a standard treatment for metastatic castrate-resistant prostate cancer (mCRPC) but treatment failure and side effects remain significant concerns. Researchers are identifying non-castrating therapies to improve treatment tolerance and quality of life. Recently, the anti-tumor effect of sodium-glucose cotransporter 2 (SGLT2) inhibitors has been revealed in vitro, vivo, and population-based observational studies. However, only one phase I trial has assessed their safety in PCa, and no randomized controlled trial (RCT) has evaluated their efficacy.

A phase 2 multicenter, open-label RCT will be performed in Queen Mary Hospital, Ruijin Hospital and Huashan Hospital (subject to Ethics Committee approval at each center) with 60 mCRPC patients proposed to be recruited. Data will be collected through radiological scan, laboratory test and case report form. Eligible patients will be randomized into two treatment groups with a 1:1 ratio. Patients in the test group will receive dapagliflozin on top of NHA plus ADT while those in the control group will receive standard of care NHA plus ADT. The primary outcome is radiographic progression-free survival. Secondary outcomes include overall survival, biomedical recurrence-free survival, time to first subsequent anti-cancer therapy, time to treatment failure, objective response rate and duration of response. Exploratory outcomes include treatment-related adverse events, quality of life, fear of cancer recurrence, and severity of pain. The primary analysis is efficacy analysis based on the intention-to-treat population. Hazard ratios will be calculated using Cox regression. Interim and finial analyses will be performed upon different study stages.

This study will be the first RCT to evaluate the efficacy and safety of SGLT2 inhibitors combined with the first-line next-generation hormonal agent (NHA) for mCRPC treatment. Given their general tolerability and clinical use, repurposing SGLT2 inhibitors as a non-castrating therapy may lead to better outcomes for PCa patients. Findings of this study will inform a novel combination therapy for advanced PCa, potentially enhancing clinical practice guidelines for its treatment and management in Hong Kong and mainland China

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years and above
* Histologically or cytologically confirmed diagnosis of prostatic adenocarcinoma without neuroendocrine/ small cell histology;
* PCa progression while receiving ADT (or post bilateral orchiectomy) within 6 months before screening: two consecutive rising PSA levels, radiographic soft tissue or bone progression;
* Current evidence of metastatic disease by radiological scan;
* Decided to receive any of the NHA (including Abiraterone Acetate, Enzalutamide, Apalutamide or Darolutamide) under standard of care setting, or started NHA for no more than 28 days at the time of treatment period start;
* Ongoing androgen deprivation with serum testosterone <50 ng/dL (<1.7 nM);
* Naïve of taxane-based chemotherapy regimens;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Normal hematologic and organ function as defined below: (a) leukocytes ≥ 3,000/mcL; (b) absolute neutrophil count ≥ 1,500/mcL; (c) platelets ≥ 100,000/mcL; (d) total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN); (e) AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN; (f) estimated glomerular filtration rate eGFR ≥ 30 mL/min/1.73m2;
* Ability to understand and willingness to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Current or previous treatment with SGLT2 inhibitors or thiazolidinedione;
* Presence of type 1 diabetes mellitus, insulin-requiring diabetes mellitus or poorly controlled diabetes mellitus (i.e., HbA1c > 10%, unless approved by endocrinologist);
* Presence of malignancies other than prostate cancer within two years prior to study enrollment;
* Disease progressed during or after treatment with one NHA;
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dapagliflozin;
* Clinically significant abnormal serum potassium or sodium level;
* Presence of uncontrolled comorbidities including but not limited to ongoing or active infection (e.g., HIV, HBV, HCV and tuberculosis), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, peripheral arterial disease, ketoacidosis, severe kidney disease, symptomatic hypotension, and chronic/frequent urinary tract infections or yeast infections;
* Participation in another clinical trial with therapeutic intent within 28 days prior to enrollment;
* Inability to swallow capsules/tablets
* Any medical conditions that might deem unsafe or contraindicated for inclusion in the clinical trial, per investigator's discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostate cancer is only available on biological male with Y chromosome
Enrollment: 60 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until the date of first disease progression per RECIST 1.1 criteria, assessed up to 60 months
  Progression free survival of prostate cancer per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of date of death from any cause, assessed up to 60 months
  Overall survival
Adverse Event | All adverse events will be evaluated once every 3 months since the date of randomization, until 1 year after the end of treatment, or resolution of any treatment related adverse event, whichever is later.
  Adverse Event of combination therapy (dapagliflozin + ADT + NHA)
Duration of response | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months.
  The time from randomization to disease progression or death, only in patients who achieve complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Yung Na, BM, MD, MPH, Principal Investigator — The University of Hong Kong
Locations (2):
- China (2):
  - Huashan Hospital, Shanghai
  - Ruijin Hospital, Shanghai